CLINICAL TRIAL: NCT01243203
Title: Smoking Cessation Program in the Preadmission Clinic: The Use of a Teachable Moment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Frances Chung, Staff Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: GA30517W
Record Dates: First submitted 2010-11-16; First posted 2010-11-18 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2013-11

CONDITIONS: Smoking
Keywords: Smoking, surgery, Anesthesia, quit
MeSH Terms: conditions — Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo (Placebo Comparator): patient will receive placebo pills
  Interventions: Drug: Champix

INTERVENTIONS:
Drug: Champix — Days 1 - 3: 0.5 mg once daily (1 table each day) Days 4 - 7: 0.5 mg twice daily (1 in the morning and 1 in the evening) Days 8 - 12 weeks 1.0 mg twice daily (1 in the morning and 1 in the evening)

SUMMARY:
The Objective of this study is to introduce a practically feasible multifaceted intervention in the preadmission clinic to help reduce smoking in preoperative surgical patients. The investigators aim to study the effectiveness of such a program in promoting positive change in smoking behavior among patients before surgery. The forced abstinence enforced on patients during hospital stay for their surgery can also be used to help smokers remain tobacco free long term. A significant percentage of surgical patients will be receptive to smoking cessation interventions in the preadmission clinic and will refrain from smoking at 24 and 52 weeks after starting the treatment.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will recruit patients who are assessed in preadmission clinic and scheduled for elective surgical procedures within the next 8 to 30 days.
* Patients should be 18 yrs of age, have smoked an average 10 cigarettes/day or more during the previous year and had no period of smoking abstinence longer than 3 months in the past year.

Exclusion Criteria:

* current pregnancy, breastfeeding;
* major depression, panic disorder, psychosis, or bipolar disorder within the prior year;
* use of nicotine replacement or bupropion within the previous 3 months;
* cardiovascular disease within the past 6 months;
* a serious or unstable disease within the past 6 months;
* drug or alcohol abuse or dependence within the past year;
* and use of tobacco products other than cigarettes or marijuana use within the previous month;
* participating in any other studies
* Patients who cannot understand English or have any form of cognitive impairment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-11; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
A significant percentage of surgical patients will be receptive to smoking cessation interventions in the preadmission clinic and will refrain from smoking at 24 and 52 weeks after starting the treatment. | 2 years

SECONDARY OUTCOMES:
Patients who receive interventions but do not quit smoking will have reduced number of cigarettes consumed /day or improved "stage of change" (determined by Prochaska and DiClemente's Model) at 24 and 52 weeks after starting the treatment. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Department of Anesthesai, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273